CLINICAL TRIAL: NCT00599612
Title: An Open Label Study to Determine the Safety, Tolerability, Excretion Balance and Pharmacokinetics of [14C]GW856553, Administered as a Single Dose of an Oral Solution to Healthy Adult Male Subjects
Brief Title: To Assess the Excretion Balance and Pharmacokinetics of a Single Oral Dose of [14C]GW856553 in Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107806
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GW856553,; radiolabel; ADME,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy male volunteers (Experimental): Six healthy male volunteers aged between 30-60 years old will be recruited for this study,
  Interventions: Drug: GW856553

INTERVENTIONS:
Drug: GW856553 — A dose of 10mg GW856553 containing 50µCi of [14C]GW856553 will be delivered as 100mL of a 0.1mg/mL GW856553/0.5 µCi/mL oral solution.

SUMMARY:
This will be an open label study conducted at one site. Six healthy male subjects will be enrolled to ensure at least four fully evaluable subjects. Each subject will receive a single 10 milligram (mg) oral dose of GW856553 containing 50 microCi (µCi) of [14C] GW856553. Urine and fecal samples will be collected until 216 hour after dosing but subjects may be discharged after 168 hour if 90% of the dose is recovered and/or <1% of the dose is excreted in a 24 hour period. Blood and plasma will be collected at various sample times after dosing to measure parent drug and total drug-related material. Samples of urine, faeces and plasma will be transferred into a separate study to characterize and quantify metabolites in these matrices. Safety will be assessed by adverse event monitoring, vital signs, electrocardiogram (ECG) and clinical laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged between 30 and 60 years inclusive, at the time of screening.
* Body weight >/ 50 kilogram (kg).
* A body mass index (BMI) within the range of 18.5 to 29.9 kg/ meter square (m^2) inclusive.
* Signed and dated written informed consent prior to admission to the study.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination, or ECG (12-lead).
* Significant cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
* QT interval corrected by Bazett's Formula (QTcB) > 450 milliseconds (msecs)
* A definite or suspected personal or family history of adverse reactions or hypersensitivity to the trial drug or to drugs with a similar chemical structure.
* History of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units). One unit is equivalent to a half-pint [284 milliliter (mL)] of beer/lager; 25mL measure of spirits or 125mL of wine).
* Subjects with a history or presence of gastro-intestinal or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Subjects who have consumed grapefruit or grapefruit juice within seven days of the first study day.
* Subjects who have had exposure to more than three new chemical entities within 12 months prior to the first dosing period.
* Subjects who have participated in a trial with a different new chemical entity within 90 days prior to the start of this study.
* If participation in the study will result in the volunteer having donated more than 400mL of blood in the previous 56 days.
* Subjects who have received a total body radiation dose of greater than 5.0 mSv (upper limit of WHO category II) or exposure to significant radiation (e.g. serial X-ray or CT scans, barium meal etc) in the 12 months prior to this study.
* History of elevated blood pressure or blood pressure persistently >140/90 mmHg at screening.
* An unwillingness to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, sub dermal implants or a tubal ligation if the women could become pregnant from the time of the first dose of the study medication until completion of the follow-up procedures.
* Lack of suitability for participation in this study, for any reason, in the opinion of the investigator.
* Any condition that could interfere with the accurate assessment and recovery of 14C.
* Prescribed or over-the-counter medication within 5 days (or 5 half lives, whichever is longer) prior to the first dosing day, unless the investigator confirms that it will not introduce additional risk or interfere with the study procedures or outcome.
* Liver function tests (ALT, AST, ALP, Gamma GT and bilirubin) > upper limit of normal (ULN) at screening
* Positive urine drug screen
* Positive HIV, Hepatitis B or C result at screening.
* History of use of tobacco- or nicotine-containing products within 6 months of screening or a positive urine cotinine screen (urine cotinine > 250ng/ml).

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01-17 (Actual); Primary Completion 2008-02-18 (Actual); Study Completion 2008-02-18 (Actual)

PRIMARY OUTCOMES:
Percentage of the total radioactive dose administered over time | Up to 10 days
  The urinary and fecal cumulative excretion will be analyzed.

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) from time zero to infinity (AUC[0-inf]) of total drug | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Blood samples will be collected at specific time points for calculating AUC (0-inf)
Maximum plasma concentration(Cmax) of total drug | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Blood samples will be collected at specific time points for calculating Cmax
AUC from zero to the time of the last measurable concentration (AUC[0-t]) of total drug | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Blood samples will be collected at specific time points for calculating AUC(0-t)
First time of occurrence of maximum observed concentration (Tmax) of total drug | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Blood samples will be collected at specific time points for calculating Tmax
Terminal plasma half-life (t1/2) of total drug | Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose
  Blood samples will be collected at specific time points for calculating T1/2
AUC(0-inf) of GW856553 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples will be collected at specific time points for calculating AUC(0-inf)
AUC(0-inf) of GSK198602 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples for metabolite analysis will be collected at specific time points for calculating AUC(0-inf)
Cmax of GW856553 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples will be collected at specific time points for calculating Cmax
Cmax of GSK198602 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples for metabolite analysis will be collected at specific time points for calculating Cmax
AUC(0-t) of GW856553 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples will be collected at specific time points for calculating AUC(0-t)
AUC(0-t) of GSK198602 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples for metabolite analysis will be collected at specific time points for calculating AUC(0-t)
Tmax of GW856553 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples will be collected at specific time points for calculating Tmax
Tmax of GSK198602 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples for metabolite analysis will be collected at specific time points for calculating Tmax
T1/2 of GW856553 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples will be collected at specific time points for calculating T1/2
T1/2 of GSK198602 | Pre-dose and 1, 4, 12 hours post-dose
  Blood samples for metabolite analysis will be collected at specific time points for calculating T1/2
Number of subjects with Adverse events (AEs) and serious adverse events (SAEs) | Up to 15 days
  An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Number of subjects with abnormal ECG findings | Up to 15 days
  Full 12-lead ECGs will be recorded using an ECG machine
Number of subjects with abnormal blood pressure values | Up to 15 days
  Systolic and diastolic blood pressure values will be measured in a supine position having rested in this position for at least 10 minutes before each reading.
Number of subjects with abnormal heart rate values | Up to 15 days
  Heart rate values will be measured in a supine position having rested in this position for at least 10 minutes before each reading.
Number of subjects with abnormal clinical chemistry parameters | Up to 15 days
  Samples for clinical chemistry tests will be collected as a measure of safety
Number of subjects with abnormal clinical hematology parameters | Up to 15 days
  Samples for clinical hematology tests will be collected as a measure of safety
Number of subjects with abnormal urine analysis parameters | Up to 15 days
  Urine samples for urine analysis tests will be collected as a measure of safety
Number of subjects with abnormal liver function tests | Up to 15 days
  Samples for liver function tests will be collected as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Edinburgh, United Kingdom